CLINICAL TRIAL: NCT03643744
Title: Photodynamic Therapy-Induced Immune Modulation: Part III
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Per PI due to data analysis results.
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06499
Record Dates: First submitted 2018-08-14; First posted 2018-08-23 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Actinic Keratosis; Photodynamic Therapy
Keywords: Actinic Keratosis; Photodynamic Therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- PDT + Celecoxib (Active Comparator): Patient receiving PDT taking 200mg celecoxib.
  Interventions: Drug: Celecoxib 200mg
- PDT + Placebo (Placebo Comparator): Patient receiving PDT taking placebo.
  Interventions: Drug: Placebo
- Control + Celecoxib (Active Comparator): Control subject not receiving PDT taking 200mg celecoxib.
  Interventions: Drug: Celecoxib 200mg
- Control + Placebo (Placebo Comparator): Control subject not receiving PDT taking placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib 200mg — 14 Celecoxib 200mg taken 1 in the morning and 1 in the evening.
  Arms: Control + Celecoxib; PDT + Celecoxib
Drug: Placebo — 14 placebo capsules taken 1 in the morning and 1 in the evening.
  Arms: Control + Placebo; PDT + Placebo

SUMMARY:
This study is designed as a double-blinded proof of concept of feasibility study to define if the immunosuppression associated with photodynamic therapy (PDT) can be blocked by treatment with cyclo-oxygenase-2 (COX-2) inhibitor celecoxib in comparison to placebo. PDT consists of application of the photosensitizer 5-aminolevulinic acid followed by treatment with a blue light. PDT is used to treat pre-cancerous actinic keratosis on large areas of skin. These studies are a continuation of ongoing studies that indicate that the lipid mediator platelet-activating factor (PAF) is generated in skin following PDT, and that PDT suppresses the immune system. It is hypothesized that PDT-generated PAF results in the immunosuppression associated with PDT. Therefore, it is proposed that a treatment to block that immunosuppression could protect the patient undergoing PDT. Blockers of the PAF system are not currently commercially available. However research studies done at Wright State University using mice indicate that PAF- and PDT-induced immunosuppression is blocked by treatment with COX-2 inhibitors. This study is conducted as a proof of concept.

Study length and visit for subjects with actinic keratoses: The first part of the study is completed in 12 days then there are follow up visits at 6 and 12 months. There are a total of 6 separate visits to the research office.

Study length and visit for control subjects: The study is completed in 10 days. There are a total of 4 separate visits to the research office.

ELIGIBILITY:
Inclusion Criteria for Control Subjects:

* Adult age 45 or older
* Caucasian (Fair skin, Fitzpatrick types I and II)
* Ability to understand and consent to the instructions of the study
* Have access to stable transportation

Inclusion Criteria for Study Subjects:

* Wright State University dermatologist has prescribed PDT for the treatment of actinic damage (Presence of precancerous actinic keratoses whose treatment necessitates PDT with the BLU-U).
* Undergoing PDT on greater than 5% body surface area: face and scalp, face and dorsal surface of arms, face and chest, face and back, or dorsal surface of arms alone, chest alone, or back alone.
* Caucasian (Fair skin, Fitzpatrick types I and II)
* Adult-age 45 or older
* Ability to understand the informed consent and comply with instructions and have stable transportation.

Exclusion Criteria for All Subjects:

* PDT on less than 5% body surface area (eg, forehead)
* Present treatment with corticosteroids or Non-steroidal inflammatory drugs (e.g., cyclooxygenase inhibitors) within past 2 months (except low-dose 81 mg aspirin).
* On antioxidant supplements (e.g., vitamin C) for past 2 months
* Tanning bed use within last 3 months
* PDT treatments within last 3 months
* Significant health issues that could affect the immune system (e.g., uncontrolled Diabetes Mellitus, Rheumatoid arthritis, skin rashes, psoriasis) that could interfere with testing
* Pregnant or nursing
* No immunosuppression, and on no immunosuppressive medications or NSAIDS within past 30 days (except low-dose [81 mg daily] aspirin).
* No significant underlying diseases that could potentially interfere with the immune assays or cardiac or renal or liver problems.
* History of blood clot or hypercoagulable state or GI bleed/ulceration.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Dayton, OH area. Patients who were prescribed to undergo photodynamic therapy (PDT) for actinic keratoses at Wright State Physicians were recruited. The control (patients who did not need photodynamic therapy) subjects where also recruited from Wright State Physicians or from the community.
Groups:
- PDT + Celecoxib: Patient receiving PDT taking 200mg celecoxib.
  Celecoxib 200mg: 14 Celecoxib 200mg taken total over 7 days (1 is taken in the morning and 1 is taken in the evening).
- PDT + Placebo: Patient receiving PDT taking placebo.
  Placebo: 14 placebo capsules taken total over 7 days (1 is taken in the morning and 1 is taken in the evening).
- Control + Celecoxib: Control subject not receiving PDT taking 200mg celecoxib.
  Celecoxib 200mg: 14 Celecoxib 200mg taken total over 7 days (1 is taken in the morning and 1 is taken in the evening).
- Control + Placebo: Control subject not receiving PDT taking placebo.
  Placebo: 14 placebo capsules taken total over 7 days (1 is taken in the morning and 1 is taken in the evening).
Period: Overall Study
Arm/Group | PDT + Celecoxib | PDT + Placebo | Control + Celecoxib | Control + Placebo
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PDT + Celecoxib | PDT + Placebo | Control + Celecoxib | Control + Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 3 | 4
  >=65 years | 3 | 3 | 2 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 4
  Male | 3 | 2 | 2 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Photodynamic Therapy (PDT)-Induced Systemic Immunosuppression From Baseline With Celecoxib Treatment.
Description: Investigator measures areas of inflammation from the reactions to intradermal (candida and trichophyton antigens) skin testing to calculate the areas of reaction. The areas of induration were measured using calipers with cm2 as the unit of measurement. The outcome measurement was calculated by using the cm2 measurements from baseline and Day 7 to calculate the percentage of initial reaction area.
Time Frame: Baseline and Day 7
Measure: Mean (Standard Error); unit: Percentage of initial reaction area
Arm/Group | PDT + Celecoxib | PDT + Placebo | Control + Celecoxib | Control + Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3
Percentage of initial reaction area | 152 (107) | 78 (19) | 206 (58) | 170 (44)
Statistical Analysis 1: Comparison: PDT + Celecoxib vs PDT + Placebo; Test type: Superiority; p = 0.530, ANOVA
Statistical Analysis 2: Comparison: Control + Celecoxib vs Control + Placebo; Test type: Superiority; p = 0.727, ANOVA

2. Primary Outcome: Change From Baseline in the Number of Actinic Keratosis at 6 Months.
Description: Investigator will assess the number of actinic keratosis in the PDT-treated areas.
Time Frame: 6 Months after PDT treatment at Day 0
Population: Study was terminated before this outcome measurement time frame occurred, therefore data was not collected for this outcome.
Arm/Group | PDT + Celecoxib | PDT + Placebo | Control + Celecoxib | Control + Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: PDT + Celecoxib vs PDT + Placebo; Test type: Superiority; p > 0.05, t-test, 2 sided

3. Primary Outcome: Change From Baseline in the Number of Actinic Keratosis at 12 Months.
Description: Investigator will assess the number of actinic keratosis in the PDT-treated areas.
Time Frame: 12 Months after PDT treatment at Day 0
Population: as for outcome 2
Arm/Group | PDT + Celecoxib | PDT + Placebo | Control + Celecoxib | Control + Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events collection started on Day -2 and ended at the end of the study (12 month follow up visit for subjects who received photodynamic therapy and at Day 11 for control subjects).
Arm/Group | PDT + Celecoxib | PDT + Placebo | Control + Celecoxib | Control + Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03643744/Prot_SAP_002.pdf
  • Informed Consent Form: Research Subjects (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03643744/ICF_000.pdf
  • Informed Consent Form: Control Subjects (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03643744/ICF_001.pdf